CLINICAL TRIAL: NCT01449682
Title: Efficacy of an Intravitreal Dexamethasone Implant on Macular Function in Retinal Vein Occlusion Following Treatment With Intravitreal Anti-VEGF Injections.
Brief Title: Efficacy of an Intravitreal DEX Implant in Retinal Vein Occlusion Following Treatment With Anti-VEGF Injections.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Retina Macula Institute (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIT-287
Record Dates: First submitted 2011-10-06; First posted 2011-10-10 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-04

CONDITIONS: Retinal Vein Occlusion; Macular Edema
Keywords: BRVO; CRVO; Macular Edema; Anti-VEGF; Ozurdex
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — Calcium Dobesilate; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ozurdex PRN (Active Comparator): 0.7 mg intravitreal DEX implant at Visit 1 then PRN for duration of trial (48 weeks) if evidence of fluid on OCT
  Interventions: Drug: Ozurdex
- Ozurdex Q16 weeks (Active Comparator): 0.7 mg intravitreal DEX implant at Visit 1 then Q16 weeks
  Interventions: Drug: Ozurdex

INTERVENTIONS:
Drug: Ozurdex — 0.7 mg intravitreal DEX implant on first visit, then PRN if evidence of macular edema on OCT studies
  Other Names: Dexamethasone implant, DEX implant
  Arms: Ozurdex PRN
Drug: Ozurdex — 0.7 mg intravitreal DEX implant on first visit then every 16 weeks
  Other Names: dexamethasone implant, DEX implant
  Arms: Ozurdex Q16 weeks

SUMMARY:
To test the efficacy of a 0.7 mg intravitreal dexamethasone implant (Ozurdex®) on macular function and recalcitrant macular edema associated with retinal vein occlusion following treatment with 2 or more prior intravitreal anti-VEGF drug injections.

DETAILED DESCRIPTION:
The efficacy of the DEX implant on macular edema for RVO is well established in multiple clinical trials. However, the duration and frequency of re-treatment have not been extensively explored. In addition, no prior studies have tested the efficacy of the DEX implant on retinal and macular function using diagnostic testing measurements such as multi-focal ERG, microperimetry and RAM testing. Since VA and OCT outcomes do not always correlate, these other assessments (mf-ERG, microperimetry, RAM testing) may be useful as early predictors of when or if patients should be retreated. This study will assess 2 groups (0.7mg PRN and 0.7mg Q16 weeks) and assess high resolution OCT, RAM testing, microperimetry, and Multi-focal ERG outcomes. For the PRN group retreated based on any fluid on OCT, we will investigate if microperimetry or multifocal ERG changes would have been an earlier predictor of fluid returning.

ELIGIBILITY:
Inclusion Criteria:

* Presence of central retinal vein occlusion (CRVO) or branch retinal vein occlusion (BRVO)
* Prior treatment with >= 2 intravitreal anti-VEGF injections but no treatment in last 45 days.
* Age 18 years or older
* ETDRS Visual acuity between 3 and 72 letters and approximate Snellen equivalent of 20/25 to 20/800
* Central foveal thickness >275 microns or presence of cystic edema on OCT studies.
* For sexually active women of childbearing potential, agreement to the use of an appropriate form of contraception (or abstinence) for the duration of the study.
* Ability to provide written informed consent • Capable of complying with study protocol

Exclusion Criteria:

* History of steroid-related glaucoma (steroid response) requiring more than one topical glaucoma medication.
* Intraocular injection of steroid medication within prior 4 months
* Evidence of significant retinal ischemia on fluorescein angiography in the opinion of the treating physician.
* Previous laser photocoagulation within 4 months of study
* Concurrent ocular disease (e.g proliferative diabetic retinopathy, geographic atrophy) that would limit visual acuity in the opinion of the treating physician
* Patients who are pregnant.
* Unwilling or unable to follow or comply with all study related procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-10; Primary Completion 2012-07 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron P Gallemore, M.D. Ph.D, Principal Investigator — Retina Macula Institute; Behnam Sharareh, B.S, Study Director — Retina Macula Institute
Locations (1):
- Retina Macula Institute, Torrance, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Comparator: Ozurdex PRN: Drug: dexamethasone intravitreal implant Ozurdex, 0.7 mg intravitreal dexamethasone implant, given at initial visit and PRN every 16 weeks
  Other Name: Ozurdex PRN
- Active Comparator: Ozurdex q16 Weeks: Drug: dexamethasone intravitreal implant Ozurdex, 0.7 mg intravitreal dexamethasone implant, given at initial visit and every 16 weeks
  Other Name: Ozurdex q16 weeks
Period: Overall Study
Arm/Group | Active Comparator: Ozurdex PRN | Active Comparator: Ozurdex q16 Weeks
Started | 5 | 5
Completed | 4 | 4
Not Completed | 1 | 1
Not completed — Death | 0 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ozurdex PRN: Drug: dexamethasone intravitreal implant Ozurdex, 0.7 mg intravitreal dexamethasone implant, given at initial visit and PRN every 16 weeks
  Other Name: Ozurdex PRN
- Ozurdex q16 Weeks: Drug: dexamethasone intravitreal implant Ozurdex, 0.7 mg intravitreal dexamethasone implant, given at initial visit and every 16 weeks
  Other Name: Ozurdex PRN
- Total: Total of all reporting groups
Arm/Group | Ozurdex PRN | Ozurdex q16 Weeks | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (5.7) | 63.3 (8.0) | 66.2 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Macular Function Using Microperimetry
Description: To determine if there is change in mean macular sensitivity using microperimetry at 48 weeks compared to baseline for both the PRN and Q16weeks treatment groups
Time Frame: baseline to 48 weeks
Measure: Mean (Standard Error); unit: dB
Arm/Group | Ozurdex PRN | Ozurdex Q16 Weeks
Number analyzed (Participants) | 5 | 5
dB
  Baseline | 2.7 (0.8) | 12.7 (2.6)
  Final Visit | 4.2 (1.7) | 10.7 (1.9)

2. Primary Outcome: Macular Function Using Multi-focal ERG
Description: To determine if there is a change in central amplitude responses using multifocal ERG at 48 weeks compared to baseline values for both the PRN and Q16weeks treatment groups
Time Frame: baseline to 48 weeks
Measure: Mean (Standard Error); unit: nV/deg2
Arm/Group | Ozurdex PRN | Ozurdex Q16 Weeks
Number analyzed (Participants) | 5 | 5
nV/deg2
  Baseline | 3.61 (0.39) | 6.62 (0.83)
  Final Visit | 18.20 (4.03) | 30.18 (9.60)

3. Secondary Outcome: To Determine if There is a Change in Visual Acuity (Number of ETDRS Letters) at 48 Weeks Compared to Baseline Values for Both the PRN and Q16weeks Treatment Groups
Time Frame: baseline to 48 weeks
Measure: Mean (Standard Error); unit: ETDRS letters
Arm/Group | Ozurdex PRN | Ozurdex Q16 Weeks
Number analyzed (Participants) | 5 | 5
ETDRS letters
  Baseline | 46.4 (7.1) | 55.6 (7.5)
  Final Visit | 27.8 (8.4) | 53.2 (8.5)

4. Secondary Outcome: To Determine if There is a Change in Central Foveal Thickness (Microns on High Resolution OCT) at 48 Weeks Compared to Baseline Values for Both the PRN and Q16weeks Treatment Groups
Time Frame: baseline to 48 weeks
Measure: Mean (Standard Error); unit: microns
Arm/Group | Ozurdex PRN | Ozurdex Q16 Weeks
Number analyzed (Participants) | 5 | 5
microns
  Baseline | 501.7 (59.7) | 353.5 (27.0)
  Final Visit | 361.4 (47.3) | 326.7 (21.2)

ADVERSE EVENTS:
Arm/Group | Ozurdex PRN | Ozurdex Q16 Weeks
All-Cause Mortality (participants affected / at risk) | 0/5 | 1/5
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ozurdex PRN (N=5) | Ozurdex Q16 Weeks (N=5)
Cataract Requiring Emergent Surgery (Eye disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ozurdex PRN (N=5) | Ozurdex Q16 Weeks (N=5)
Elevated Intraocular Pressure (Eye disorders) | 0 (0) | 1 (1) — Greater than 10 mmHg above baseline measure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No